CLINICAL TRIAL: NCT04534868
Title: Evaluation of Patients Acceptance and Satisfaction With Teledermoscopy at the General Practionner's Office for the Detection of Skin Cancer in a Rural Area.
Brief Title: Patient Acceptance And Satisfaction of Teledermoscopy In General Practice In a Belgian Rural Area
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CE 2020/06AOU/397
Record Dates: First submitted 2020-08-17; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Skin Cancer; Patient Acceptance of Health Care; Patient Satisfaction
Keywords: Skin Cancer Screening; General Practice; Teledermoscopy; Patient Satisfaction and Acceptance
MeSH Terms: conditions — Skin Neoplasms; Patient Acceptance of Health Care; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Acceptance and satisfaction for teledermoscopy (Other): The aim of the first part of the study is to evaluate patients' skin monitoring habits, their knowledge of skin cancer, and their preconceptions about new telemedicine tools such as teledermoscopy. This is a written quantitative questionnaire with answers to tick.
  An explanatory folder will be given to patients and they will be asked to read it beforehand in order to allow a good understanding of the terms used and the goal of the project. This part will include 70 to 100 patients.
  The second part of the study is a qualitative study and the aim of it is to evaluate the satisfaction, acceptance and future expectations of those who have benefited from teledermoscopy. Individual and anonymous interviews, lasting 15 to 20 minutes, intended for patients who have benefit of teledermoscopy at the office. An explanatory folder will also be given to the patients concerned in order to explain to them the procedure of the interview. This part will include 8 to 10 patients.
  Interventions: Other: taking macroscopic and dermoscopic pictures of suspicious skin lesions

INTERVENTIONS:
Other: taking macroscopic and dermoscopic pictures of suspicious skin lesions — If there is any diagnostic doubt about a skin lesion, teledermoscopy will be used, if the patient agrees.
  * A table containing the useful information about the patient for the lesion's analysis will be completed.
  * The pictures will be taken with a Fotofinder Handyscope. The photos will be integrated into the patient's electronic medical record (CareConnect program).
  * The photo is anonymized via a serial number assigned by the "Handyscope" application.
  * Sending photos and information via a secure email address to the dermatologists.
  * Response from the dermatologist (Prof. Tromme or Dr Harkemanne) in the following days also via email.
  * Contact (consultation or telephone call depending on the diagnosis) with the patient to communicate the results and the procedure to be followed.
  * This information (emails containing the dermatological report) will be saved in the patient's computerized medical file (CareConnect program) then deleted from the mailbox

SUMMARY:
The aim objective of this work is to assess the characteristics of patients for whom teledermoscopy could be suitable for the detection of potential skin cancers, within a population of rural general medicine in the South of Hainaut, by means of a mixed quantitative and qualitative study corresponding respectively:

* To identify patients' knowledge of skin cancers, their skin monitoring habits, and their acceptability of new telemedicine tools such as teledermoscopy ("Part 1").
* To evaluate the satisfaction and expectations of those who benefit from teledermoscopy ("Part 2").

ELIGIBILITY:
Inclusion Criteria:

* Adults ( > 18y)
* French Speaking Patient

Exclusion Criteria:

* Illiterate Patients
* Demented Patients
* Non-French speaking patients
* Minors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-03-15 (Estimated)

PRIMARY OUTCOMES:
Patient Acceptability Of Teledermoscopy | 20 to 30 minutes to complete the questionnaire.
  Using a quantitative survey-type questionnaire
  * Determination of the patients ' skin monitoring habits
  * Determination of patients' knowledge of skin cancers and their prevention
  * Determine their acceptance of new technologies such as teledermoscopy in the context of skin cancer screening
  * And finally, determination of a target population for whom teledermoscopy could be suitable for the detection of skin cancers (percentage of patients accepting teledermoscopy etc)
Patient Satisfaction after a teledermoscopy experience | 15 to 20 minutes (interview duration)
  Assessment of the satisfaction and future expectations of patients who have benefited from teledermoscopy in general practice, using a qualitative study in the form of semi-structured, individual and anonymous interviews

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tensen E, van der Heijden JP, Jaspers MW, Witkamp L. Two Decades of Teledermatology: Current Status and Integration in National Healthcare Systems. Curr Dermatol Rep. 2016;5:96-104. doi: 10.1007/s13671-016-0136-7. Epub 2016 Mar 28. PMID 27182461
- [Background] Kips J, Lambert J, Ongenae K, De Sutter A, Verhaeghe E. Teledermatology in Belgium: a pilot study. Acta Clin Belg. 2020 Apr;75(2):116-122. doi: 10.1080/17843286.2018.1561812. Epub 2019 Jan 8. PMID 30618351
- [Background] Tan E, Yung A, Jameson M, Oakley A, Rademaker M. Successful triage of patients referred to a skin lesion clinic using teledermoscopy (IMAGE IT trial). Br J Dermatol. 2010 Apr;162(4):803-11. doi: 10.1111/j.1365-2133.2010.09673.x. Epub 2010 Mar 5. PMID 20222920
- [Background] Borve A, Dahlen Gyllencreutz J, Terstappen K, Johansson Backman E, Aldenbratt A, Danielsson M, Gillstedt M, Sandberg C, Paoli J. Smartphone teledermoscopy referrals: a novel process for improved triage of skin cancer patients. Acta Derm Venereol. 2015 Feb;95(2):186-90. doi: 10.2340/00015555-1906. PMID 24923283
- [Background] van Sinderen F, Tensen E, van der Heijden JP, Witkamp L, Jaspers MWM, Peute LWP. Is Teledermoscopy Improving General Practitioner Skin Cancer Care? Stud Health Technol Inform. 2019 Aug 21;264:1795-1796. doi: 10.3233/SHTI190652. PMID 31438348
- [Background] Vestergaard T, Prasad SC, Schuster A, Laurinaviciene R, Bygum A, Munck A, Andersen MK. Introducing teledermoscopy of possible skin cancers in general practice in Southern Denmark. Fam Pract. 2020 Sep 5;37(4):513-518. doi: 10.1093/fampra/cmaa041. PMID 32347299
- [Background] Koh U, Horsham C, Soyer HP, Loescher LJ, Gillespie N, Vagenas D, Janda M. Consumer Acceptance and Expectations of a Mobile Health Application to Photograph Skin Lesions for Early Detection of Melanoma. Dermatology. 2019;235(1):4-10. doi: 10.1159/000493728. Epub 2018 Nov 7. PMID 30404081
- [Background] Kong F, Horsham C, Rayner J, Simunovic M, O'Hara M, Soyer HP, Janda M. Consumer Preferences for Skin Cancer Screening Using Mobile Teledermoscopy: A Qualitative Study. Dermatology. 2020;236(2):97-104. doi: 10.1159/000505620. Epub 2020 Mar 3. PMID 32126557
- [Background] Snoswell CL, Whitty JA, Caffery LJ, Loescher LJ, Gillespie N, Janda M. Direct-to-consumer mobile teledermoscopy for skin cancer screening: Preliminary results demonstrating willingness-to-pay in Australia. J Telemed Telecare. 2018 Dec;24(10):683-689. doi: 10.1177/1357633X18799582. PMID 30343653
- [Background] Hue L, Makhloufi S, Sall N'Diaye P, Blanchet-Bardon C, Sulimovic L, Pomykala F, Colomb M, Baccard M, Lassau F, Reuter G, Keller F, Fite C, Triller R, Cremieux AC. Real-time mobile teledermoscopy for skin cancer screening targeting an agricultural population: an experiment on 289 patients in France. J Eur Acad Dermatol Venereol. 2016 Jan;30(1):20-4. doi: 10.1111/jdv.13404. Epub 2015 Nov 16. PMID 26568080
- [Background] Damsin T, Jacquemin P, Canivet G, Giet D, Gillet P, Nikkels AF. [TeleSPOT Project : early detection of melanoma by teledermoscopy in general practice]. Rev Med Liege. 2019 Dec;74(12):650-654. French. PMID 31833275
- [Background] Gilling S, Mortz CG, Vestergaard T. Patient Satisfaction and Expectations Regarding Mobile Teledermoscopy in General Practice for Diagnosis of Non-melanoma Skin Cancer and Malignant Melanoma. Acta Derm Venereol. 2020 Apr 21;100(8):adv00117. doi: 10.2340/00015555-3459. PMID 32179927
- [Background] Mounessa JS, Chapman S, Braunberger T, Qin R, Lipoff JB, Dellavalle RP, Dunnick CA. A systematic review of satisfaction with teledermatology. J Telemed Telecare. 2018 May;24(4):263-270. doi: 10.1177/1357633X17696587. Epub 2017 Mar 28. PMID 28350281
- [Background] Kruse CS, Krowski N, Rodriguez B, Tran L, Vela J, Brooks M. Telehealth and patient satisfaction: a systematic review and narrative analysis. BMJ Open. 2017 Aug 3;7(8):e016242. doi: 10.1136/bmjopen-2017-016242. PMID 28775188
- See also: Related Info — https://www.agoria.be/fr/Le-coronavirus-active-le-remboursement-de-la-tele-consultation